CLINICAL TRIAL: NCT00226187
Title: A Randomized Clinical Trial on Supplementation of DHA and AA to Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2005-09-22; First posted 2005-09-26 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2005-09

CONDITIONS: Infant, Low Birth Weight
Keywords: Fatty acids; Human milk; Infant development; Very low birthweight infants

INTERVENTIONS:
Procedure: Supplement of fatty acid (DHA and AA)

SUMMARY:
A randomized, double-blind trial of docosahexaenoic and arachidonic acid supplementation in breast-fed preterm infants

Background:

Docosahexaenoic acid (DHA) and arachidonic acid (AA) are essential for preterm infants. Human milk and preterm formulas contain DHA and AA, but at lower concentrations than required to approximate utero accretion rate.

Objective:

To evaluate the effect of a high dose DHA and AA supplement to breast-fed preterm infants in the early neonatal period. Primary endpoints are neurodevelopment at 6 and 20 months of age.

Design:

A randomized double-blind placebo-controlled study is carried out in four Norwegian neonatal centers.

Subjects and methods:

Infants with birth weight < 1.5 kg are randomized to either an intervention or a control group. All infants receive fortified human milk, and a daily dose of 0.5 ml study oil per 100 ml milk. Infants in the intervention group receive oil with DHA and AA (Formulaid, Martek, USA), while the control oil contains vegetable oil without DHA or AA. Blood samples are collected at birth (cord), and at start and stop of the intervention. Plasma is analyzed for fatty acid pattern using high performance liquid chromatography.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight < 1500 g
* Born at one of 4 participating neonatal centers in Norway

Exclusion Criteria:

* Cerebral haemorrhage (stage 3 or 4)
* Major congenital malformations that are supposed to affect growth and development
* Illness that require prolonged parenteral nutrition (>4 weeks)

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140
Dates: Start 2003-12

PRIMARY OUTCOMES:
Cognitive development

SECONDARY OUTCOMES:
Growth
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Christian A Drevon, Dr. Med., Study Chair — University og Oslo
Locations (1):
- University of Oslo, Oslo, Oslo County, Norway

REFERENCES:
- [Derived] Almaas AN, Tamnes CK, Nakstad B, Henriksen C, Grydeland H, Walhovd KB, Fjell AM, Iversen PO, Drevon CA. Diffusion tensor imaging and behavior in premature infants at 8 years of age, a randomized controlled trial with long-chain polyunsaturated fatty acids. Early Hum Dev. 2016 Apr;95:41-6. doi: 10.1016/j.earlhumdev.2016.01.021. Epub 2016 Mar 2. PMID 26939082
- [Derived] Almaas AN, Tamnes CK, Nakstad B, Henriksen C, Walhovd KB, Fjell AM, Due-Tonnessen P, Drevon CA, Iversen PO. Long-chain polyunsaturated fatty acids and cognition in VLBW infants at 8 years: an RCT. Pediatrics. 2015 Jun;135(6):972-80. doi: 10.1542/peds.2014-4094. Epub 2015 May 18. PMID 25986018
- [Derived] Henriksen C, Haugholt K, Lindgren M, Aurvag AK, Ronnestad A, Gronn M, Solberg R, Moen A, Nakstad B, Berge RK, Smith L, Iversen PO, Drevon CA. Improved cognitive development among preterm infants attributable to early supplementation of human milk with docosahexaenoic acid and arachidonic acid. Pediatrics. 2008 Jun;121(6):1137-45. doi: 10.1542/peds.2007-1511. PMID 18519483